CLINICAL TRIAL: NCT01088152
Title: Structured Education of Swedish Celiac Women Living on a Gluten-free Diet for Years
Brief Title: Celiac Disease School for Women Living on a Gluten-free Diet
Acronym: CDST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Research Council of Southeast Sweden (Other Government)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Norrkoping Hospital, Claes HallertMD PhD, Norrkoping Hospital, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORSS-80731; M218-08 (Other: Ethics Committee at Linkoping University, Linkoping Sweden)
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2001-01

CONDITIONS: Education of Patients; Counseling; Problem-Based Learning
Keywords: Celiac disease; Education; Sweden; Gluten-free diet
MeSH Terms: conditions — Celiac Disease | interventions — Patient Education as Topic; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care of celiac disease women (Active Comparator): Written information corresponding to that offered when seeking medical advice for celiac disease in primary care
  Interventions: Behavioral: Usual care of celiac disease women
- Celiac School (Experimental): Structured education using problem-based learning at 10 sessions
  Interventions: Behavioral: Celiac school

INTERVENTIONS:
Behavioral: Celiac school — Structured education of adult celiac patients at 10 sessions.
  Other Names: Patient education; Counselling
  Arms: Celiac School
Behavioral: Usual care of celiac disease women — Written information corresponding to that offered when seeking medical advice for well treated celiac disease in the primary care.
  Other Names: Coeliac disease guidelines
  Arms: Usual care of celiac disease women

SUMMARY:
Swedish celiac disease women living on a gluten-free diet for years report poorer subjective health and more bowel complaints than Swedish women of same age in general population.

The investigators hypothesis is that the women participating in an education programme based on problem based learning will show higher degree of perceived health than the women receiving usual care.

DETAILED DESCRIPTION:
Celiac disease is a disorder of the small intestines triggered by dietary gluten, a protein in wheat-containing foods. Living with is far from easy and associated with restrictions and various dilemmas in daily life, leading to depressed mood and reduced well-being, particularly in women. We decided to include 100 celiac disease women on a gluten-free diet into a randomized controlled education trial in order to compare problem-based learning with usual care. Outcome measures will be two frequently employed questionnaires: PGWB (Psychological Well-being Index) to monitor Well-being and GSRS (Gastrointestinal Symptom Rating Scale) to measure the rate bowel symptoms as assessed at 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 yrs or above with Celiac disease treated for at least five years

Exclusion Criteria:

* Anticipated inability to comply the trial protocol

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Subjective health and well-being | 6 months
  Gastrointestinal symptoms and Psychological well-being

SECONDARY OUTCOMES:
Gastrointestinal symptoms and Psychological well-being | 6 months
  Two questionnaires: Psychological General Well-Being Index and the Gastrointestinal Symptom Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Claes Hallert, MD, PhD, Study Director — Norrkoping Hospitalö
Locations (1):
- Norrkoping Hospital,, Norrköping, Sweden

REFERENCES:
- [Background] Hallert C, Sandlund O, Broqvist M. Perceptions of health-related quality of life of men and women living with coeliac disease. Scand J Caring Sci. 2003 Sep;17(3):301-7. doi: 10.1046/j.1471-6712.2003.00228.x. PMID 12919466
- [Background] Sverker A, Hensing G, Hallert C. 'Controlled by food'- lived experiences of coeliac disease. J Hum Nutr Diet. 2005 Jun;18(3):171-80. doi: 10.1111/j.1365-277X.2005.00591.x. PMID 15882379
- [Background] Midhagen G, Hallert C. High rate of gastrointestinal symptoms in celiac patients living on a gluten-free diet: controlled study. Am J Gastroenterol. 2003 Sep;98(9):2023-6. doi: 10.1111/j.1572-0241.2003.07632.x. PMID 14499782
- [Background] Roos S, Karner A, Hallert C. Psychological well-being of adult coeliac patients treated for 10 years. Dig Liver Dis. 2006 Mar;38(3):177-80. doi: 10.1016/j.dld.2006.01.004. Epub 2006 Feb 7. PMID 16461026